CLINICAL TRIAL: NCT05592145
Title: Quantifying the Venous Congestion Curve of a Tissue Oximetry Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB00090046
Record Dates: First submitted 2022-10-19; First posted 2022-10-24 (Actual); Results first posted 2024-03-20 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2023-10

CONDITIONS: Post-Op Complication; Skin Flap Necrosis
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Intervention Model Description: The ViOptix machine will be used to measure the oxygenation of composite tissue.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- ViOptix T.Ox (Other): ViOptix T.Ox machine is used to measure the oxygenation of composite tissue.
  Interventions: Device: ViOptix

INTERVENTIONS:
Device: ViOptix — ViOptix machine

SUMMARY:
The purpose of this research study is to measure rate of decline and pattern of tissue oxygenation using the device, ViOptix T.Ox.

ViOptix probes will be secured to the arm and hand. The recording process on the ViOptix machine will begin and obtain baseline StO2 levels for 5 minutes. After 5 minutes, a blood pressure cuff will be inflated on one arm. This blood pressure cuff will be left inflated for 10-20 minutes. Every 2 minutes a pulse check or doppler exam will be performed at your wrist. Last, the cuff will be deflated and the you will be free to leave the study room.

DETAILED DESCRIPTION:
The rate of decline and pattern seen in tissue oxygenation as quantified by a NIRS device (ViOptiox T.Ox) can be quantified and described by a mathematical model which will allow earlier detection and identification of venous congestion in tissue. The vascular occlusion test has been established as a safe and accurate model to induce various states of vascular insufficiency and occlusion. Specifically the vascular occlusion test has been demonstrated to be an accurate model for inducing venous insufficiency on awake and aware patients. This study will aim to analyze the StO2 data output of the ViOptix in order to establish the earliest signs of tissue failure in various states of vascular compromise.

The purpose of this research study is to measure rate of decline and pattern of tissue oxygenation using the device, ViOptix T.Ox. The data collected will be used to formulate a mathematical model which will allow earlier detection and identification of venous congestion in tissue. Identifying these specific patterns will help to establish an evidence-based approach in recognizing specific problems and patterns associated with tissue compromise that can guide physicians to consider earlier flap salvage measures.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 65 volunteers

Exclusion Criteria:

* Subjects with a history of major cardiac disease, peripheral vascular disease including (vascular insufficiency), Raynaud syndrome, blood dyscrasias, pain syndromes, neurologic conditions, major upper extremity soft tissue trauma or previous vascular injury

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2022-11-10 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ramon Llull, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ViOptix T.Ox
Started | 38
Completed | 38
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | ViOptix T.Ox
Number analyzed (Participants) | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 38
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 25.5 [22 to 37]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 38

OUTCOME MEASURES:

1. Primary Outcome: Transcutaneous Oximetry (StO2) of Vascular Occlusion Test at 0.5 Hours
Description: transcutaneous oximetry (StO2) of vascular occlusion test at 0.5 hours - an StO2 greater than 55 mmHg is considered normal regardless of the site of measurement
Time Frame: Hour 0.5
Measure: Mean (Full Range); unit: percentage of oxygen saturation
Arm/Group | ViOptix T.Ox
Number analyzed (Participants) | 38
percentage of oxygen saturation | 70.353 [0 to 100]

ADVERSE EVENTS:
Time Frame: Each participant was in the study and monitored for adverse events for approximately one hour on the day the study activities occurred.
Arm/Group | ViOptix T.Ox
All-Cause Mortality (participants affected / at risk) | 0/38
Serious Adverse Events (participants affected / at risk) | 0/38
Other Adverse Events (participants affected / at risk) | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-10-27): https://cdn.clinicaltrials.gov/large-docs/45/NCT05592145/Prot_SAP_001.pdf
  • Informed Consent Form (2023-10-26): https://cdn.clinicaltrials.gov/large-docs/45/NCT05592145/ICF_000.pdf